CLINICAL TRIAL: NCT00004051
Title: A Phase I Study to Evaluate Orally Administered Irinotecan HCL (CPT-11) Given as a Powder-Filled Capsule Formulation Daily for 14 Days Every Three Weeks in Patients With Advanced Solid Tumors
Brief Title: Irinotecan in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067246; MSKCC-98076; P-UPJOHN-976475155; NCI-G99-1569
Record Dates: First submitted 1999-12-10; First posted 2004-05-20 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2009-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of irinotecan in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose, dose limiting toxicity, and safety profile of oral irinotecan in patients with advanced solid tumors. II. Characterize the single and multiple dose pharmacokinetics of oral irinotecan and its metabolites, SN-38 and SN-38 glucuronide, in these patients. III. Document any antitumor activity in these patients treated with this regimen.

OUTLINE: This is a dose escalation study. Patients receive oral irinotecan once daily for 14 days. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 or more of 6 patients experience dose limiting toxicity. Patients are followed monthly for 6 months.

PROJECTED ACCRUAL: Approximately 3-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced solid tumor for which no curative therapy exists No leukemias or lymphomas Brain or leptomeningeal disease allowed only if prior irradiation of these lesions, no concurrent corticosteroids, and no clinical symptoms

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 150,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL regardless of liver tumor presence SGOT no greater than 3 times upper limit of normal (ULN) (5 times ULN if due to liver tumor) Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No uncontrolled high blood pressure No unstable angina No symptomatic congestive heart failure No myocardial infarction within past 6 months No serious uncontrolled cardiac arrhythmia Gastrointestinal: No active inflammatory bowel disease No significant bowel obstruction No chronic malabsorption Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active infection HIV negative No AIDS related illness No significant alcoholism or substance abuse No severe medical or psychiatric illness that would preclude participation in study

PRIOR CONCURRENT THERAPY: At least 4 weeks since prior therapy for cancer and recovered Biologic therapy: No concurrent immunotherapy No concurrent filgrastim (G-CSF), sargramostim (GM-CSF), or epoetin alfa Chemotherapy: No prior nitrosoureas, mitomycin, or irinotecan No prior high dose chemotherapy in support of peripheral blood stem cell transplantation No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: No prior irradiation of pelvis No concurrent radiotherapy Surgery: No prior gastrectomy or total colectomy Other: At least 1 week since prior anticonvulsants No other concurrent investigational drugs No combination anticholinergic medications containing barbiturates (e.g., Donnatol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1998-08; Primary Completion 2001-07 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States